CLINICAL TRIAL: NCT03839134
Title: The Effectiveness of Automated Soft Tissue Vibration in Reducing Pain and Accelerating Action of Intraoral Local Anesthesia Injections in Adult Dental Patients. A Randomized Crossover Clinical Trial.
Brief Title: The Effectiveness of Soft Tissue Vibration in Reducing Pain of Local Anesthesia Injection in Adult Dental Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Ra'ed Salma, Assistant Professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: FRP/2018/286
Record Dates: First submitted 2019-01-30; First posted 2019-02-15 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Anesthetics, Local
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Pain of buccal injection with DentalVibe® (Experimental): DentalVibe® Comfort Injection System will be used prior and during the local anesthesia (LA) buccal injection. The LA to be used is Lidocaine 2% with Epinephrine dental injection.
  Interventions: Device: DentalVibe® Comfort Injection System; Drug: Lidocaine Epinephrine
- Pain of buccal injection without DentalVibe® (Active Comparator): Local anesthesia (LA) for buccal infiltration using Lidocaine Epinephrine dental injection. No tissue vibrations will be performed before or during the injection.
  Interventions: Drug: Lidocaine Epinephrine
- Pain of palatal injection with DentalVibe® (Experimental): DentalVibe® Comfort Injection System will be used prior and during the local anesthesia (LA) palatal injection. The LA to be used is Lidocaine 2% with Epinephrine dental injection.
  Interventions: Device: DentalVibe® Comfort Injection System; Drug: Lidocaine Epinephrine
- Pain of palatal injection without DentalVibe® (Active Comparator): Local anesthesia (LA) for palatal infiltration using Lidocaine Epinephrine dental injection. No tissue vibrations will be performed before or during the injection.
  Interventions: Drug: Lidocaine Epinephrine
- Pain of block injection with DentalVibe® (Experimental): DentalVibe® Comfort Injection System will be used prior and during the local anesthesia (LA) injection for inferior alveolar nerve (IAN) block. The LA to be used is Lidocaine 2% with Epinephrine dental injection.
  Interventions: Device: DentalVibe® Comfort Injection System; Drug: Lidocaine Epinephrine
- Pain of block injection without DentalVibe® (Active Comparator): Local anesthesia (LA) injection for inferior alveolar nerve (IAN) block using Lidocaine Epinephrine dental injection. No tissue vibrations will be performed before or during the injection.
  Interventions: Drug: Lidocaine Epinephrine

INTERVENTIONS:
Device: DentalVibe® Comfort Injection System — Soft tissue vibration for 10 seconds using DentalVibe®. The device induces approximately 16 soft tissue vibrations of per second. The device will be in touch of oral mucosa (at the site of injection) before and during the local anesthesia injection.
  Other Names: DentalVibe
  Arms: Pain of block injection with DentalVibe®; Pain of buccal injection with DentalVibe®; Pain of palatal injection with DentalVibe®
Drug: Lidocaine Epinephrine — Dental local anesthesia injection of 1.8 mL Lidocaine (2%) with Epinephrine (1:80000 w/v).
  Other Names: Xylocaine 2% with Epinephrine

SUMMARY:
The clinical trial will compare pain perception during dental local anesthesia injections with and without using soft tissue vibration device prior to injection. The primary goal is to test the effectiveness of such devices in pain/discomfort reduction during intraoral local anesthesia injections in various techniques (infiltration and block anesthesia).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status class I
* Planned for multiple dental treatments in the maxilla and mandible bilaterally

Exclusion Criteria:

* Patients <18 years old
* Pregnant ladies
* Smokers and alcoholics
* Patients on medications
* Drug abusers
* Never received dental treatment under local anesthesia before
* Patients with an acute infection with or without fever
* Patients with preoperative pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Pain of needle penetration of buccal LA injection | 1-2 seconds after mucosal penetration
  The pain of needle penetration will be assessed using 10-point Graphic Rating Scale (GRS). The pain score will be compared to its counterpart pain score on the experimental side using DentalVibe® injection system.
Pain of anesthesia delivery during buccal LA infiltration | 30 seconds after LA solution delivery
  The pain during anesthesia solution delivery will be assessed using 10-point Graphic Rating Scale (GRS). The pain score will be compared to its counterpart pain score on the experimental side using DentalVibe® injection system.
Pain of needle penetration of palatal LA injection | 1-2 seconds after mucosal penetration
  The pain of needle penetration will be assessed using 10-point Graphic Rating Scale (GRS). The pain score will be compared to its counterpart pain score on the experimental side using DentalVibe® injection system.
Pain of anesthesia delivery during palatal LA infiltration | 30 seconds after LA solution delivery
  The pain during anesthesia solution delivery will be assessed using 10-point Graphic Rating Scale (GRS). The pain score will be compared to its counterpart pain score on the experimental side using DentalVibe® injection system.
Pain of needle penetration of IAN block LA injection | 1-2 seconds after mucosal penetration
  The pain of needle penetration will be assessed using 10-point Graphic Rating Scale (GRS). The pain score will be compared to its counterpart pain score on the experimental side using DentalVibe® injection system.
Pain of anesthesia delivery during IAN block LA injection | 30 seconds after LA solution delivery
  The pain during anesthesia solution delivery will be assessed using 10-point Graphic Rating Scale (GRS). The pain score will be compared to its counterpart pain score on the experimental side using DentalVibe® injection system.

CONTACTS AND LOCATIONS:
Overall Officials: Ra'ed G Salma, Principal Investigator — Riyadh Elm University
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No